CLINICAL TRIAL: NCT04076761
Title: A Multi-Centre, Open-Label Phase 2 Study of TRIFLURIDINE/TIPIRACIL in Previously Treated Cholangiocarcinoma (The MOCHA Trial)
Brief Title: Study of TRIFLURIDINE/TIPIRACIL in Previously Treated Cholangiocarcinoma
Acronym: MOCHA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO 1645
Record Dates: First submitted 2019-08-22; First posted 2019-09-03 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Cholangiocarcinoma; Bile Duct Cancer
Keywords: Cholangiocarcinoma; Bile Duct Cancer; FTD/TPI; TRIFLURIDINE/TIPIRACIL
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trifluridine/Tipiracil (Experimental): FTD/TPI at 35 mg/m2 (based on BSA) that is administered in tablet form, orally, twice daily, within one hour of morning and evening meals, on days 1-5 and days 8-12 of a 28 day cycle.
  Interventions: Drug: Trifluridine/Tipiracil

INTERVENTIONS:
Drug: Trifluridine/Tipiracil — FTD/TPI is an orally administered combination of a thymidine-based nucleic acid analogue, trifluridine, and a thymidine phosphorylase inhibitor, tipiracil hydrochloride. Trifluridine is the active cytotoxic component of FTD/TPI; its triphosphate form is incorporated into DNA, with such incorporation appearing to result in its anti- tumor effects. Tipiracil hydrochloride is a potent inhibitor of thymidine phosphorylase and, when combined with trifluridine to form FTD/TPI, prevents the rapid degradation of the trifluridine, allowing for the maintenance of adequate plasma levels of the active drug.
  Other Names: FTD/TPI; Lonsurf

SUMMARY:
This is a multi-centre, open-label, single arm phase 2 study to assess the efficacy of TRIFLURIDINE/TIPIRACIL, in patients with advanced cholangiocarcinoma as measured by median progression-free survival (PFS).

This study will enroll a total of 47 patients over a 12-month period, according to a two stage enrollment design. Nine patients will be enrolled during the first stage and the trial will be terminated if 4 or more out of the 9 have disease progression. If the trial goes on to the second stage, a total of 47 patients (38 in second stage) will be required.

Patients will be seen prior to enrolment (within 28 days of treatment), every 4 weeks while on treatment, at the end of treatment, and 30 days post-treatment. Patients will remain on long-term follow-up and will be seen every 12 weeks (+/- 14 days) until 1 year post-treatment when they will enter into the survival follow-up period and will be contacted every 12 weeks by phone until progression or toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented locally advanced or metastatic biliary tract cancer (intra or extrahepatic cholangiocarcinoma or gallbladder cancer) previously treated with first line standard chemotherapy (gemcitabine-based chemotherapy at least one cycle). Patients who develop a recurrence after adjuvant capecitabine therapy must have subsequently received at least one cycle of a gemcitabine-based therapy to be eligible. Patients who have received gemcitabine in the adjuvant setting but progressed within 6 months of their last cycle will be eligible for the study.
2. Presence of measurable disease as assessed by CT scan of the chest, abdomen and pelvis based on RECIST 1.1.
3. ECOG performance status of 0 or 1.
4. Expected life expectancy of ≥ 3 months.
5. Age 18 years and above
6. Able to swallow and retain oral medication.
7. Adequate hematologic function defined by the following laboratory parameter:

   1. Hemoglobin ≥ 9g/dL
   2. Absolute neutrophil count ≥1.5 x 109/L
   3. Platelet count ≥75x 109/L
8. Adequate hepatic and renal function as defined by:

   1. AST and ALT ≤ 3.0 X ULN (≤ 5 if liver metastasis present)
   2. Total bilirubin ≤ 1.5X ULN
   3. Calculated creatinine clearance ≥50 ml/min using Cockcroft-Gault formula
9. Patients who have treated brain metastasis (via local radiation standards or surgical resection or local techniques) and who are either off steroids or on a stable dose of steroids for at least one month (30 days), AND who are off anticonvulsants, AND have radiological documented stability of lesions for at least 3 months may be eligible.
10. Patients must have the ability to read, understand, and sign an informed consent and must be willing to comply with study treatment and procedures.

Exclusion Criteria:

1. Any malignancy related to HIV, history of HIV, history of known HBV surface antigen positivity (subjects with documented laboratory evidence of HBV clearance may be enrolled) or positive HCV antibody. Testing for these diseases is not mandatory unless clinically indicated
2. Chemotherapy, radiotherapy, immunotherapy, or other anti-cancer therapy including investigational drugs within 28 days prior to enrolment.
3. Patients with unresolved Grade 3/4 toxicities from prior therapies.
4. Any major surgery within the last four weeks.
5. Previous or concurrent malignancies, excluding curatively treated in situ carcinoma of the cervix or uterus or non-melanoma skin cancer or in-situ carcinoma of the prostate (Gleason score ≤ 7, with all treatment being completed 6 months prior to enrollment, unless at least 5 years have elapsed since last treatment and the patient is considered cured)
6. Patients with locally or centrally known FGFR2 fusion (Sunnybrook, Ottawa and PMCC sites only).
7. Female patients of childbearing potential and men able to father children who do not agree to use adequate methods of contraception from time of enrolment until 6 months after the last date of treatment administration.
8. Women who are breastfeeding
9. Patients with suspected or documented leptomeningeal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Median progression-free survival (PFS) | From enrolment until the date of objective radiological disease progression according to RECIST v1.1 or death (by any cause in the absence of progression) up to 1 year
  As measured on the basis of RECIST v1.1 criteria

SECONDARY OUTCOMES:
Safety and tolerability of FTD/TPI: CTCAE version 5.0 | Day 1 of each new treatment cycle (each cycle is 28 days), and at the end of treatment visit (up to 1 year after enrolment)
  Assessed by using CTCAE version 5.0 and tolerability
Disease Control Rate (Complete Response, Partial Response, Stable Disease) of FTD/TPI | From enrolment until the date of objective radiological disease progression according to RECIST v1.1 or death (by any cause in the absence of progression) up to 1 year
  As measured on the basis of RECIST v1.1 criteria
Duration of response of FTD/TPI | From enrolment until the date of objective radiological disease progression according to RECIST v1.1 or death (by any cause in the absence of progression) up to 1 year
  As measured on the basis of RECIST v1.1 criteria
Median overall survival of patients with cholangiocarcinoma treated with FTD/TPI. | From enrolment until the date of objective radiological disease progression according to RECIST v1.1 or death (by any cause in the absence of progression) up to 1 year
  As measured on the basis of RECIST v1.1 criteria
Quality of life: European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 | Baseline, and Day 1 of each new treatment cycle (each cycle is 28 days), and at the end of treatment visit (up to 1 year after enrolment)
  As measured by the European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC-QLQ C30) Functioning, symptoms, and global health status scores will be calculated, graphed, and summarized at baseline and each follow-up visit. General linear mixed model will be conducted to detect significant changing over time for functioning, symptoms and global health status scores. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada